CLINICAL TRIAL: NCT04196712
Title: Essen Coronary Artery Disease Registry
Acronym: ECAD registry
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-8956-BO
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Coronary angiography arm: Patient undergoing invasive coronary angiography

SUMMARY:
The ECAD registry is a registry of patients undergoing coronary angiography at the West German Heart and Vascular Center. The registry anticipates to determine predictors of patient outcome after coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing invasive coronary angiography at the West German Heart and Vascular Center

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This registry includes all consecutive patients undergoing invasive coronary angiography at the West German Heart and Vascular Center, starting from 2003.
Sampling Method: Non-Probability Sample
Enrollment: 55000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | through study completion, an average of 3 year
  Mortality of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, Principal Investigator — University Hospital Essen, Deparment of Cardiology and Vascular Medicine
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No